CLINICAL TRIAL: NCT03319212
Title: Clinical Characterization of Symptomatic Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5969
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active Comparator (Other): Subjects that are between the ages 18-55 and are current spherical soft contact lens wearers will be assigned to a single study lens type to be worn bilaterally for approximately 4 weeks followed by no contact lens wear for 1 week.
  Interventions: Device: senofilcon A contact lenses

INTERVENTIONS:
Device: senofilcon A contact lenses — Senofilcon A Daily Disposable Contact Lenses

SUMMARY:
This is an unmasked, non-randomized, single arm, stratified, dispensing investigation of symptomatic and asymptomatic subject populations. Subjects will be assigned to a single study lens type to be worn bilaterally for approximately 4 weeks followed by no contact lens wear for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 55 (inclusive) years of age at the time of screening.
  4. Be a current soft contact lens wearer in both eyes with a minimum of 3 days/week wear time over the last 1 month by self-report.
  5. Have a baseline CLDEQ-8 score of either:

     1. 7 or lower
     2. 15 or greater
  6. Subjects must possess a functional / usable pair of spectacles and bring them to the visit (only if applicable - to the investigators discretion).
  7. Subjects must pass a pre-screening questionnaire.
  8. Subjects must be willing to discontinue all contact lens wear for approximately 1 week/
  9. Subjects must present to visit 1 with their habitual lenses on eye for at least 6 hours.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating, by self-report.
  2. Any ocular or systemic allergies, disease or use of medication which may interfere with contact lens wear (at the discretion of the investigator).
  3. Any active ocular abnormalities/conditions that may interfere with contact lens wear (at the discretion of the investigator).
  4. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
  5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
  6. Habitual contact lens wear modality as extended wear (≥1 night per month of extended wear).
  7. Habitual contact lens is rigid gas permeable, toric, monovision or multi-focal
  8. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
  9. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
  10. Employee or employee's immediate family member of clinical site (e.g., Investigator, Coordinator, Technician).
  11. Current habitual use of Restasis, Xiidra, ocular steroids, or any medication (RX or OTC) that may interfere with contact lens wear (at the discretion of the investigator).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- VRC-East, Jacksonville, Florida, United States
- University of Waterloo Center for Contact Lens Research, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 105 subjects were enrolled into this study. Of those enrolled 81, were dispensed a study lens while 24 subjects failed to meet all eligibility criteria. Of those dispensed a study lens, 73 completed the study while 8 subjects were discontinued. All subjects were disepsned the same study lens senofilcon A.
Pre-assignment Details: Subjects were stratified into two subject groups: symptomatic (baseline CLDEQ-8 score of 15 or greater) and asymptomatic (baseline CLDEQ-8 score of 7 or lower).
Groups:
- Asymptomatic: Subjects with baseline CLDEQ-8 score of 7 or lower were assigned to the asymptomatic group throughout the entire duration of the study. All subjects wore the senofilcon A lens in both eyes throughout the entire duration.
- Symptomatic: Subjects with baseline CLDEQ-8 score of 15 or greater were assigned to the symptomatic group throughout the entire duration of the study. All subjects wore the senofilcon A lens in both eyes throughout the entire duration.
Period: Overall Study
Arm/Group | Asymptomatic | Symptomatic
Started | 29 | 52
Completed | 26 | 47
Not Completed | 3 | 5
Not completed — Discontinued as moving out of local area | 0 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asymptomatic: Subjects with baseline CLDEQ-8 score of 7 or lower were assigned to the asymptomatic group throughout the entire duration of the study
- Symptomatic: Subjects with baseline CLDEQ-8 score of 15 or greater were assigned to the symptomatic group throughout the entire duration of the study.
- Total: Total of all reporting groups
Arm/Group | Asymptomatic | Symptomatic | Total
Number analyzed (Participants) | 29 | 52 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.76 (7.229) | 28.17 (9.096) | 28.38 (8.4333)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 36 | 54
  Male | 11 | 16 | 27
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 7 | 20 | 27
  Black or African American | 1 | 2 | 3
  White | 21 | 27 | 48
  Other | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 14 | 25
  Canada | 18 | 38 | 56

OUTCOME MEASURES:

1. Primary Outcome: Meibomian Gland Imaging
Description: Meibomian gland imaging was assessed in each each subject eye, at baseline, 4-Week Follow-up (during lens wear) and the the 5-Week Follow-up on subjects' bare eyes. Meibomian gland imaging is expressed interms of area of loss using the following grading scale: Degree 0 ≈ 0%; Degree 1 ≤ 25%; Degree 2 26% - 50%; Degree 3 51% - 75%; Degree 4 ≥ 75%.
Time Frame: 4-Week Follow-up
Population: All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hardlock.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
eyes
  Degree 0 | 10 | 4
  Degree 1 | 23 | 66
  Degree 2 | 18 | 16
  Degree 3 | 1 | 8

2. Primary Outcome: Meibomian Gland Expressibility
Description: Meibomian glands were assessed in the three regions of each lower eyelid: temporal, central, and nasal. Approximately five glands are expressed per region with each use of the Meibomian Gland Evaluator. Secretions for each of the 5 glands selected within the three regions were graded using the following secretion grading scale: Grade 0 = No Secretion (Includes capped orifices), Grade 1 = Inspissated (semi-solid, toothpaste-like consistency), Grade 2 = Colored/Cloudy Liquid, Grade 3 = Clear Liquid Oil. The total grades for 5 glands per region was calculated for each subject. The total Meibomian Gland Secretion Score was calculated by adding the grades for the 15 glands assessed. Mean and standard deviation for total grade per region and total Meibomian Gland Secretion Score were reported for each stratum. Total scores range from 0 to 15 were lower score indicate worsening meibomian gland expressability.
Time Frame: 4-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
Score on a Scale
  Central Lower Lid | 9.04 (5.068) | 8.07 (5.055)
  Temporal Lower Lid | 8.71 (4.795) | 7.94 (4.803)
  Nasal Lower Lid | 7.94 (4.976) | 6.54 (4.571)
  Total Score | 25.69 (13.964) | 22.55 (12.649)

3. Primary Outcome: Lid Margin Evaluation: Number of Eyes With Abnormal Biomicroscopy Findings
Description: Lid margin evaluation was conducted for upper and lower lids for both left and right eyes. The presence of the following biomicroscopy findings were recorded as No/normal or Yes/abnormal:
  * Irregularity: Notching of Margin
  * Vascularity of Lid Margin: Telangiectasia
  * Meibomian Gland Pouting, Plugging, or Capping
  * Lid/Lash Margin Debris Findings.
  The number of positive findings (yes) was reported for each group.
Time Frame: 4-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
Number of eyes
  Irregularity: Notching of Margin | 1 | 5
  Vascularity of Lid Margin: Telangiectasia | 12 | 21
  Meibomian Gland Pouting, Plugging, or Capping | 12 | 33
  Lid/Lash Margin Debris Findings | 0 | 10

4. Primary Outcome: Lid Wiper Epitheliopathy
Description: Horizontal length of staining and sagittal width of staining were graded for both upper and lower lids for each eye. Average grade was calculated separately for upper and lower lids, and the final grade was calculated as the average grade across upper and lower lids. Mean and standard deviation were reported for the final grade by stratum. Subjects were classified according to their final lid wiper epitheliopathy grade for each eye using the following scale: None = 0, Mild = 0.25 - 1.00, Moderate = 1.25 - 2.00, and Severe = 2.25 - 3.00. Final Grades range from 0 to 3, where higher final grades indicate worsening lid wiper epitheliopathy.
Time Frame: 4-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
Units on a scale | 0.50 (0.718) | 0.28 (0.489)

5. Primary Outcome: Conjunctival Folds
Description: Lid-parallel conjunctival folds (LIPCOF) will be evaluated in the area perpendicular to the temporal and nasal limbus on the bulbar conjunctiva above the lower lid (temporal and nasal LIPCOF, respectively), and classified using the LIPCOF grading scale: 0 = No conjunctival folds, 1 = One permanent and clear parallel fold, 2 = Two permanent and clear parallel folds (normally lower than 0.2mm), and 3 = More than two permanent and clear parallel folds (normally higher than 0.2mm).
Time Frame: 4-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
eyes
  Temporal- Grade 0 | 27 | 45
  Temporal- Grade 1 | 22 | 41
  Temporal- Grade 2 | 3 | 8
  Temporal- Grade 3 | 0 | 0
  Nasal- Grade 0 | 43 | 55
  Nasal- Grade 1 | 9 | 30
  Nasal- Grade 2 | 0 | 9
  Nasal- Grade 3 | 0 | 0

6. Secondary Outcome: Conjunctival Redness
Description: Limbal and bulbar conjunctival redness were assessed or each quadrant (nasal, temporal, inferior, superior) using the following scale: 0 = Normal, 1 = Trace, 2 = Mild, 3 = Moderate, and 4 = Severe.
Time Frame: 4-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 27 | 48
Number analyzed (Eyes) | 54 | 96
eyes
  Bulbar-Nasal- Grade 0 | 12 | 11
  Bulbar-Nasal- Grade 1 | 36 | 72
  Bulbar-Nasal- Grade 2 | 6 | 13
  Bulbar-Nasal- Grade 3 | 0 | 0
  Bulbar-Nasal- Grade 4 | 0 | 0
  Bulbar-Temporal- Grade 0 | 13 | 12
  Bulbar-Temporal- Grade 1 | 37 | 73
  Bulbar-Temporal- Grade 2 | 4 | 11
  Bulbar-Temporal- Grade 3 | 0 | 0
  Bulbar-Temporal- Grade 4 | 0 | 0
  Bulbar-Inferior-Grade 0 | 23 | 27
  Bulbar-Inferior-Grade 1 | 31 | 66
  Bulbar-Inferior-Grade 2 | 0 | 3
  Bulbar-Inferior-Grade 3 | 0 | 0
  Bulbar-Inferior-Grade 4 | 0 | 0
  Bulbar-Superior- Grade 0 | 23 | 31
  Bulbar-Superior- Grade 1 | 30 | 57
  Bulbar-Superior- Grade 2 | 1 | 8
  Bulbar-Superior- Grade 3 | 0 | 0
  Bulbar-Superior- Grade 4 | 0 | 0
  Limbal-Nasal- Grade 0 | 26 | 28
  Limbal-Nasal- Grade 1 | 25 | 66
  Limbal-Nasal- Grade 2 | 3 | 2
  Limbal-Nasal- Grade 3 | 0 | 0
  Limbal-Nasal- Grade 4 | 0 | 0
  Limbal-Temporal- Grade 0 | 24 | 33
  Limbal-Temporal- Grade 1 | 28 | 58
  Limbal-Temporal- Grade 2 | 2 | 5
  Limbal-Temporal- Grade 3 | 0 | 0
  Limbal-Temporal- Grade 4 | 0 | 0
  Limbal-Inferior- Grade 0 | 27 | 40
  Limbal-Inferior- Grade 1 | 27 | 55
  Limbal-Inferior- Grade 2 | 0 | 1
  Limbal-Inferior- Grade 3 | 0 | 0
  Limbal-Inferior- Grade 4 | 0 | 0
  Limbal-Superior- Grade 0 | 25 | 46
  Limbal-Superior- Grade 1 | 29 | 45
  Limbal-Superior- Grade 2 | 0 | 5
  Limbal-Superior- Grade 3 | 0 | 0
  Limbal-Superior- Grade 4 | 0 | 0

7. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining was assessed for each eye by quadrant (Superior, Inferior, Nasal, Temporal) utilizing the following scale: Grade 0 = None (No conjunctival staining), Grade 1 = Trace (Scattered superficial punctate staining), Grade 2 = Mild (Regional or generalized punctate staining), Grade 3 = Moderate (Significant coalesced punctate staining), Grade 4 = Severe (Patch staining).
Time Frame: 4-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 27 | 48
Number analyzed (Eyes) | 54 | 96
eyes
  Nasal- Grade 0 | 17 | 17
  Nasal- Grade 1 | 18 | 51
  Nasal- Grade 2 | 19 | 28
  Nasal- Grade 3 | 0 | 0
  Temporal- Grade 0 | 20 | 29
  Temporal- Grade 1 | 19 | 51
  Temporal- Grade 2 | 15 | 16
  Temporal- Grade 3 | 0 | 0
  Inferior-Grade 0 | 26 | 30
  Inferior-Grade 1 | 9 | 51
  Inferior-Grade 2 | 19 | 13
  Inferior-Grade 3 | 0 | 2
  Superior- Grade 0 | 28 | 50
  Superior- Grade 1 | 18 | 44
  Superior- Grade 2 | 8 | 2
  Superior- Grade 3 | 0 | 0

8. Secondary Outcome: Corneal Staining
Description: Corneal staining was assessed for each eye by region (Central, Superior, Inferior, Nasal, Temporal). Corneal staining type was evaluated using the following the scale: Grade 0 = None, Grade 1 = Micropunctate, Grade 2 = Macropunctate, Grade 3 = Coalesced Macropunctate, and Grade 4 = Patch (>1mm). Corneal staining area was evaluated using the following the scale: Grade 0 = 0% of region covered, Grade 1 = 10% of region covered, Grade 2 = 20% of region covered, Grade 3 = 30% of region covered, Grade 4 = 40% of region covered, Grade 5 = 50% of region covered, Grade 6 = 60% of region covered, Grade 7 = 70% of region covered, Grade 8 = 80% of region covered, Grade 9 = 90% of region covered, and Grade 10 = 100% of region covered. The following scale was used in the grading of corneal staining depth: Grade 0 = None, Grade 0 = Superficial epithelial, Grade 2 = Full epithelial, and Grade 3 = Stromal glow.
Time Frame: 4-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 27 | 48
Number analyzed (Eyes) | 54 | 96
eyes
  Staining Type- Central- Grade 0 | 51 | 88
  Staining Type- Central- Grade 1 | 1 | 5
  Staining Type- Central- Grade 2 | 2 | 3
  Staining Type- Central- Grade 3 | 0 | 0
  Staining Type-Inferior - Grade 0 | 48 | 75
  Staining Type-Inferior - Grade 1 | 5 | 17
  Staining Type-Inferior - Grade 2 | 1 | 4
  Staining Type-Inferior - Grade 3 | 0 | 0
  Staining Type-Nasal - Grade 0 | 49 | 92
  Staining Type-Nasal - Grade 1 | 4 | 2
  Staining Type-Nasal - Grade 2 | 1 | 2
  Staining Type-Nasal - Grade 3 | 0 | 0
  Staining Type-Temporal-Grade 0 | 51 | 92
  Staining Type-Temporal-Grade 1 | 2 | 2
  Staining Type-Temporal-Grade 2 | 1 | 2
  Staining Type-Temporal-Grade 3 | 0 | 0
  Staining Type- Superior- Grade 0 | 50 | 88
  Staining Type- Superior- Grade 1 | 4 | 6
  Staining Type- Superior- Grade 2 | 0 | 2
  Staining Type- Superior- Grade 3 | 0 | 0
  Staining- Area- Central- Grade 0 | 51 | 89
  Staining- Area- Central- Grade 1 | 1 | 4
  Staining- Area- Central- Grade 2 | 1 | 2
  Staining- Area- Central- Grade 3 | 1 | 1
  Staining- Area- Central- Grade 4 | 0 | 0
  Staining- Area- Central- Grade 5 | 0 | 0
  Staining- Area- Central- Grade 6 | 0 | 0
  Staining- Area- Inferior- Grade 0 | 48 | 76
  Staining- Area- Inferior- Grade 1 | 3 | 10
  Staining- Area- Inferior- Grade 2 | 0 | 8
  Staining- Area- Inferior- Grade 3 | 3 | 2
  Staining- Area- Inferior- Grade 4 | 0 | 0
  Staining- Area- Inferior- Grade 5 | 0 | 0
  Staining- Area- Inferior- Grade 6 | 0 | 0
  Staining- Area-Nasal-Grade 0 | 49 | 93
  Staining- Area-Nasal-Grade 1 | 4 | 2
  Staining- Area-Nasal-Grade 2 | 1 | 1
  Staining- Area-Nasal-Grade 3 | 0 | 0
  Staining- Area-Nasal-Grade 4 | 0 | 0
  Staining- Area-Nasal-Grade 5 | 0 | 0
  Staining- Area-Nasal-Grade 6 | 0 | 0
  Staining-Area-Temporal-Grade 0 | 51 | 92
  Staining-Area-Temporal-Grade 1 | 1 | 2
  Staining-Area-Temporal-Grade 2 | 2 | 2
  Staining-Area-Temporal-Grade 3 | 0 | 0
  Staining-Area-Temporal-Grade 4 | 0 | 0
  Staining-Area-Temporal-Grade 5 | 0 | 0
  Staining-Area-Temporal-Grade 6 | 0 | 0
  Staining-Area-Superior-Grade 0 | 50 | 89
  Staining-Area-Superior-Grade 1 | 3 | 4
  Staining-Area-Superior-Grade 2 | 0 | 3
  Staining-Area-Superior-Grade 3 | 0 | 0
  Staining-Area-Superior-Grade 4 | 1 | 0
  Staining-Area-Superior-Grade 5 | 0 | 0
  Staining-Area-Superior-Grade 6 | 0 | 0
  Staining-Depth-Central-Grade 0 | 51 | 89
  Staining-Depth-Central-Grade 1 | 3 | 7
  Staining-Depth-Central-Grade 2 | 0 | 0
  Staining-Depth-Inferior-Grade 0 | 48 | 77
  Staining-Depth-Inferior-Grade 1 | 6 | 19
  Staining-Depth-Inferior-Grade 2 | 0 | 0
  Staining-Depth-Nasal-Grade 0 | 49 | 93
  Staining-Depth-Nasal-Grade 1 | 5 | 3
  Staining-Depth-Nasal-Grade 2 | 0 | 0
  Staining-Depth-Temporal-Grade 0 | 51 | 93
  Staining-Depth-Temporal-Grade 1 | 3 | 3
  Staining-Depth-Temporal-Grade 2 | 0 | 0
  Staining-Depth-Superior-Grade 0 | 50 | 89
  Staining-Depth-Superior-Grade 1 | 4 | 7
  Staining-Depth-Superior-Grade 2 | 0 | 0

9. Secondary Outcome: Tear Film Lipid Layer Thickness
Description: Tear film lipid layer thickness was measured for each eye using LipiView II. The Review Lipid Images screen provided numerical analysis of the measured lipid layer thickness in nanometers (nm) from 10 (thinnest) to 240 (thickest), with a precision of 1 nm and an accuracy of 10 nm.
Time Frame: 4-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nm
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
nm | 66.81 (19.336) | 63.00 (16.208)

10. Secondary Outcome: Tear Film Stability
Description: Non-invasive tear break-up time (NIBUT) was measured for each eye to indicate the stability of the tear film. NIBUT is measured as the time interval in seconds after the final blink to the first appearance of distortion in the reflected rings; or to the time that the participant has to blink due to discomfort. Three measurements were taken on each eye. The average NIBUT was reported for each group.
Time Frame: 4-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
seconds | 8.03 (3.846) | 6.78 (4.327)

11. Secondary Outcome: Tear Film Lipid Pattern
Description: Tear film lipid pattern was recorded for each eye using the following categories: None, Open Meshwork, Closed (Tight Meshwork), Flow (Wave), Amorphous, Colors, and Other.
Time Frame: 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 26 | 47
Number analyzed (Eyes) | 52 | 94
eyes
  None | 0 | 0
  Open Meshwork | 6 | 24
  Closed (Tight) | 18 | 22
  Flow (Wave) | 14 | 28
  Amorphous | 11 | 15
  Colors | 3 | 5
  Others | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 5 weeks per subject.
Groups:
- Senofilcon A: All subjects that wore the senofilcon A lens at any point throughout the study.
Arm/Group | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03319212/Prot_SAP_000.pdf